CLINICAL TRIAL: NCT01234064
Title: Graduated Compression Stockings (GCS) for Prevention of Venous Thromboembolism in Patients Who Have Major Surgery: Pilot Study Assessing Feasibility of Adding This Evaluation to the PeriOperative ISchemic Evaluation-2 Trial (POISE-2 Trial)
Brief Title: Graduated Compression Stockings (GCS) Pilot Substudy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: BSN Medical Inc (Industry); McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: GCS Pilot Substudy
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2011-12

CONDITIONS: Venous Thromboembolism
Keywords: Symptomatic Venous Thromboembolism; Graduated Compression Stockings; Randomized Controlled Trial; Noncardiac Surgery
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Graduated Compression Stockings (Active Comparator)
  Interventions: Device: Anti-Embolism Graduated Pressure Stockings (by BSN-Jobst)
- No Graduated Compression Stockings (Other)
  Interventions: Device: No Graduated Compression Stockings

INTERVENTIONS:
Device: Anti-Embolism Graduated Pressure Stockings (by BSN-Jobst) — Apply 2 to 4 hours prior to surgery. Patient will continue to wear stockings until post-op Day 10.
  Other Names: Anti-Em/GP
  Arms: Graduated Compression Stockings
Device: No Graduated Compression Stockings — No stockings will be applied.
  Arms: No Graduated Compression Stockings

SUMMARY:
This is a pilot substudy to the PeriOperative ISchemic Evaluation-2 Trial (POISE-2), to assess the feasibility of adding graduated compression stockings (GCS) to POISE-2 as an intervention.

DETAILED DESCRIPTION:
Objective: To determine if thigh-level graduated compression stockings (below-knee graduated compression stockings may be used if thigh level graduated compression stockings are not feasible, such as after knee surgery), started before surgery and worn until discharge and for a minimum of 10 days (whichever is longer), reduce symptomatic venous thromboembolism (proximal deep vein thrombosis or pulmonary embolism) in the 30 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Randomized to PeriOperative ISchemic Evaluation-2 Trial (POISE-2 Trial)

Exclusion Criteria:

* Unable to wear a graduated compression stockings on a leg that has been operated on (e.g., below knee skin grafting)
* Leg has not been operated on and graduated compression stockings cannot be worn on either leg (e.g. bilateral leg amputations or skin ulceration, allergy to material in the graduated compression stockings)
* Graduated compression stockings cannot be fitted because the patient's legs are too big, or too small (not compatible with manufacturer's recommendations)
* The responsible physician/nurse judges that graduated compression stockings are contraindicated because of: i) decreased circulation in the legs as evidenced by very pale, cyanotic, or gangrenous conditions; or ii) risk of stocking-induced skin necrosis due to an established sensory neuropathy with numbness to touch.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Objectively confirmed symptomatic major venous thromboembolism | 30 days
  The primary outcome to assess efficacy will be a comparison of the proportion of patients who have objectively confirmed symptomatic major venous thromboembolism (defined as proximal deep vein thrombosis or pulmonary embolism) within 30 days of randomization (includes episodes that are diagnosed in response to symptoms reported at the 30 day assessment).

SECONDARY OUTCOMES:
Any symptomatic venous thromboembolism or pulmonary embolism | 30 days
  Secondary outcomes to assess efficacy will include patients who, within 30 days, have any symptomatic venous thromboembolism (defined as deep vein thrombosis [including that which is confined to the calf veins] or pulmonary embolism) within 30 days of randomization.
Major venous thromboembolism and death | 30 Days
  Secondary outcomes to assess efficacy will include patients who, within 30 days, have major venous thromboembolism and death.
Safety Outcomes | 30 Days
  Harm from graduated compression stockings will be assessed as proportion of patients who develop: 1) a new or worsening skin rash that required new, or an increase of, topical or systemic treatment; 2) blistering (defined as at least one blister >1cm in length); 3) pressure sores (minimum of non-blanchable erythema of intact skin); and 4) leg or foot ischaemia (defined as new symptoms (cold, painful, numbness) or new signs (pulseless, cold, absent skin perfusion on release of pressure, absent sensation) that are attributed to ischaemia by a physician.

CONTACTS AND LOCATIONS:
Overall Officials: Clive Kearon, MB, PhD, Principal Investigator — McMaster University
Locations (1):
- Henderson Hospital, Hamilton, Ontario, Canada